CLINICAL TRIAL: NCT00380757
Title: Comparison of Bystander Fatigue and CPR Quality When Using the New 30:2 Versus the Old 15:2 Chest Compression to Ventilation International Guidelines: A Randomised Crossover Trial
Brief Title: Comparison of Bystander Fatigue and CPR Quality When Using Two Different CPR Ratios.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2006347-01H
Record Dates: First submitted 2006-09-23; First posted 2006-09-26 (Estimated); Results first posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Cardiac Arrest
Keywords: cardiac arrest; CPR; resuscitation; fatigue; quality
MeSH Terms: conditions — Heart Arrest; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CPR 30:2 (Active Comparator): 30 chest compressions to 2 ventilations
  Interventions: Procedure: bystander CPR using 30:2 ratio vs 15:2 ratio
- CPR 15:2 (Active Comparator): 15 chest compressions to 2 ventilations
  Interventions: Procedure: bystander CPR using 30:2 ratio vs 15:2 ratio

INTERVENTIONS:
Procedure: bystander CPR using 30:2 ratio vs 15:2 ratio — Participants will use 2 CPR techniques with different chest compression to ventilation ratios

SUMMARY:
STUDY OBJECTIVES The overall goal of this study is to compare bystander fatigue and CPR quality after 5 minutes of the new 30:2 versus the old 15:2 chest compression to ventilation International Resuscitation Guidelines, in a population aged 55 or greater.

More specifically, we will compare each CPR ratio with regard to:

1. The achieved frequency and depth of chest compressions,
2. Participant rating of their perceived level of exertion, and
3. Resulting serum lactate levels in a subset of the participants.

STUDY HYPOTHESIS

In a population aged 55 or greater, the new 30:2 CPR ratio will lead to:

1. less frequent and shallower chest compressions over the 5-minute study period;
2. higher rating of perceived level of exertion; and
3. higher serum lactate levels in a subset of participants when compared to the old 15:2 CPR ratio.

DETAILED DESCRIPTION:
Background: Cardiac arrest is the number one cause of mortality in the Canadian population. Out-of-hospital bystander cardiopulmonary resuscitation (CPR) is associated with a 3 to 4 fold increase in survival for cardiac arrest. Any interruption in the delivery of chest compressions to cardiac arrest victims is detrimental on survival. In an effort to minimize interruptions in chest compressions, the new International Guidelines changed the long-recommended 15:2 compression to ventilation ratio to 30:2. Although the 30:2 ratio is meant to increase survival for cardiac arrest, the ability of rescuers to deliver the new CPR ratio intervention has never been studied. Little is known about the potential impact of the new recommendations on bystander fatigue and resulting CPR quality.

Objectives: The overall goal of this study is to compare bystander fatigue and CPR quality after 5 minutes of the new 30:2 versus the old 15:2 chest compression to ventilation International Guidelines in a population aged 55 or greater.

More specifically, we will compare each CPR ratio with regard to:

1. The achieved frequency and depth of chest compressions,
2. Participant rating of their perceived level of exertion, and
3. Resulting serum lactate levels in a subset of the participants.

Methods: We will conduct a randomized cross-over trial comparing bystander fatigue and CPR quality using two different CPR ratios. Intervention: All participants will be asked to perform two 5-minute sessions of CPR on a recording manikin - one session using the 30:2 ratio, the other using the 15:2 ratio. There will be a supervised practice session in the beginning, and resting periods in between. The order in which the sessions will be executed will be determined in a random fashion. The study population will consist of volunteers aged 55 or older, a group most susceptible to perform CPR on a real victim. The study will take place in a busy public area of The Ottawa Hospital, Civic Campus, between the cafeteria and the emergency department. Participants will have to score 3 or less on the validated Clinical Frailty Scale in order to participate in the study. Participants with physical limitations or disease processes precluding their ability to safely perform CPR will be excluded. Outcome measures: Information on age, gender, height, weight, prior CPR training, and measure of frailty will be collected at the time of enrollment. The number, frequency, and quality of chest compressions (depth and release) will be measured during each CPR session using a recording ResusciAnne manikin. Heart rate and blood pressure will be measured before and after each CPR sessions. The participants will be asked to rate their level of fatigue before and after each CPR session using the validated Borg Rating of Perceived Exertion scale. In addition, serum lactate levels will be determined before and after each CPR session in volunteers from the second group. Sample size: We hope to recruit 42 participants, among which 10 will have their lactate levels measured. Data analysis for Objective#1 and #3 will include descriptive statistics and a paired t-test with 95% confidence interval; Objective#2 will be analyzed using descriptive statistics and WIlcoxon Rank Sum test. In addition, we will perform a stepwise logistic regression analysis to control for the potential confounding effects of variables otherwise associated with bystander fatigue and CPR performance using both CPR ratio. This study protocol will receive ascent form the OHREB before implementation, and will be entered on the OHRI randomized trial registry.

Importance of the study Data from this study will evaluate bystander fatigue and resulting CPR quality when comparing the new 30:2 to the old 15:2 International Guidelines. This highly innovative project will improve our understanding of the physiological demands associated with the implementation of the new CPR International Guidelines. We anticipated the results from this study will be widely distributed, and will help shape the next iteration of the International Resuscitation Guidelines.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 55 or older
2. Must score 3 or less on the validated Clinical Frailty Scale 11
3. Able to follow instructions in English or French
4. Able to understand and give informed consent

   Exclusion Criteria:
5. Musculoskeletal condition precluding the ability to kneel down and perform CPR (e.g. severe arthritis, cast, wrist sprain, recent joint surgery)
6. Cardiovascular condition precluding the ability to perform a moderate effort e.g. myocardial infarction or cardiovascular procedure in the last 3 months, recurrent angina, chest pain under investigation)
7. Pulmonary condition precluding the ability to perform a moderate effort (e.g. emphysema, severe asthma, pneumonia)
8. Active communicable disease e.g. tuberculosis, meningitis, gastro enteritis, hepatitis A or B, herpes simplex)
9. Inability to perform chest compressions at appropriate rate and depth despite positive feedback during one to two-minute practice session

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2006-06 (Actual); Primary Completion 2006-07 (Actual); Study Completion 2006-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christian Vaillancourt, MD, Msc,, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- The Ottawa Hospital, Civic Campus, Ottawa, Ontario, Canada

REFERENCES:
- [Result] Vaillancourt C, Midzic I, Taljaard M, Chisamore B. Performer fatigue and CPR quality comparing 30:2 to 15:2 compression to ventilation ratios in older bystanders: A randomized crossover trial. Resuscitation. 2011 Jan;82(1):51-6. doi: 10.1016/j.resuscitation.2010.09.003. Epub 2010 Oct 14. PMID 20947241

RESULTS

PARTICIPANT FLOW:
Groups:
- CPR 30:2 First Then 15:2: 30 chest compressions to 2 ventilations
  bystander CPR using 30:2 ratio for a 5-minute period. After a 5-minute rest period, the participants will administer bystander CPR using a 15:2 ratio for 5 minutes
- CPR 15:2 First Then 30:2: 15 chest compressions to 2 ventilations
  bystander CPR using 15:2 ratio for 5 minutes, followed by a 5-minute rest period. Then participants assigned to this group will administer bystander CPR using 30:2 ratio for 5 minutes.
Period: Sequence 1 (First Assigned CPR Ratio)
Arm/Group | CPR 30:2 First Then 15:2 | CPR 15:2 First Then 30:2
Started | 21 | 21
Completed | 21 | 21
Not Completed | 0 | 0
Period: Sequence 2 (Second Assigned CPR Ratio)
Arm/Group | CPR 30:2 First Then 15:2 | CPR 15:2 First Then 30:2
Started | 21 | 21
Completed | 21 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CPR 30:2 | CPR 15:2 | Total
Number analyzed (Participants) | 21 | 21 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.4 (8.7) | 65.6 (7.1) | 66.0 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 12 | 29
  Male | 4 | 9 | 13
Region of Enrollment [Number; unit: participants]
  Canada | 21 | 21 | 42

OUTCOME MEASURES:

1. Primary Outcome: CPR Quality
Description: Number of adequate chest compressions per minute
Time Frame: over a 5 minute period
Population: Two recordings were later determined to be technically inadequate. Results are only reported for the CPR sequence that the participant was assigned to start with.
Measure: Mean (Standard Deviation); unit: count of chest compressions
Arm/Group | CPR 30:2 | CPR 15:2
Number analyzed (Participants) | 19 | 19
count of chest compressions | 128.5 (130.4) | 126.6 (129.9)

2. Secondary Outcome: Borg Rating of Perceived Exertion Blood Pressure Borg Rating of Perceived Exertion Scale
Description: Measures of bystander fatigue measured using the Borg's Scale for Rating of Perceived Exertion (range 6-20) measured at baseline, following first CPR sequence, before beginning second sequence and at end of second CPR sequence. Lower values represent light perceived exertion, and higher values represent higher perceived exertion. Values reported are the difference between the baseline Borg Scale measured before beginning each CPR sequence and the Borg Scale following 5 minutes of each CPR sequence.
Time Frame: After 5 minutes of 15:2 CPR or 30:2 CPR
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- CPR 15:2 Ratio: Mean change from baseline in Borg Rating after 5 minutes of 15:2
- CPR 30:2 Ratio: Mean change in Borg Rating from baseline after performing 5 minutes of CPR using 30:2 ratio
Arm/Group | CPR 15:2 Ratio | CPR 30:2 Ratio
Number analyzed (Participants) | 42 | 42
units on a scale | 3.3 (2.2) | 3.5 (1.9)

ADVERSE EVENTS:
Time Frame: Over the 30-min study period duration. There was no subsequent follow-up following study completion.
Arm/Group | CPR 15:2 | CPR 30:2
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/42
Other Adverse Events (participants affected / at risk) | 0/42 | 0/42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes